CLINICAL TRIAL: NCT01265979
Title: Whole Body Diffusion-weighted MRI (WB-DWI) for Early Prediction and Evaluation of Therapy Response in Patients With Advanced Metastatic Gastrointestinal Stromal Tumors (GIST) Treated With Regorafenib.
Brief Title: WB-DWI for Early Prediction of Therapy Response in Patients With Advanced Metastatic GIST Treated With Regorafenib
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, katrijn Michielsen, PhD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S52989
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: advanced; metastatic; gastro-intestinal; stromal; GIST; regorafenib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GIST treated with regorafenib/placebo: patients with advanced, metastatic gastro-intestinal stromal tumors treated with regorafenib or placebo
  Interventions: Procedure: Whole body diffusion MRI

INTERVENTIONS:
Procedure: Whole body diffusion MRI — These studies will be performed on a 3 Tesla (T) MR system. A major advantage of 3T compared to 1.5T is the improved signal to noise ratio that allows whole-body studies to be faster and without application of external antennas, which greatly improves patient comfort.

SUMMARY:
The purpose of this study is to evaluate WB DWI as early predictor of response to treatment with regorafenib or placebo in patients with advanced metastatic GIST.

DETAILED DESCRIPTION:
Aim of the study

- To assess whole body diffusion-weighted magnetic resonance imaging (WB-DWI) for the assessment and early prediction of response of treatment with regorafenib or placebo in patients with advanced, metastatic gastro-intestinal stromal tumors (GIST)

1. Evaluation of pretreatment apparent diffusion coefficient (ADC) and b1000 signal intensity (SI) of GIST visualized on the WB-DWI as predictor of time to progression, determined by progression-free survival (PFS)
2. Evaluation of WB-DWI using changes of high b-value SI and ADC early during treatment (2weeks after start of therapy; allowed optimal window 10-14 days) as early predictor of time to progression or patient benefit according to RECIST (stable disease + partial response + complete response)
3. Evaluation of WB-DWI for treatment follow-up 3 months after initiation of treatment. Confirmation of prior published pilot study (Dunet V et al, J Nucl Med 2010)
4. Comparison of WB-DWI with conventional CT imaging for response assessment

ELIGIBILITY:
Inclusion Criteria:

* patients with advanced, metastatic gastro-intestinal stromal tumors treated with regorafenib or placebo

Exclusion Criteria:

* in case of a known contraindication for MRI (eg. pacemaker), the patient will not be admitted to the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with advanced, metastatic gastro-intestinal stromal tumors treated with regorafenib or placebo
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
WB-DWI as early predictor for regorafenib treatment response | jan 2011-dec 2011
  Primary aim of the study:
  To assess whole body diffusion-weighted magnetic resonance imaging (WB-DWI) for the assessment and early prediction of response of treatment with regorafenib or placebo in patients with advanced, metastatic gastro-intestinal stromal tumors (GIST)

SECONDARY OUTCOMES:
Evaluation WB-DWI parameters in correlation with progression free survival (PFS) | jan 2011-dec 2011
  Evaluation of
  * pretreatment apparent diffusion coefficient (ADC) and b1000 signal intensity (SI)
  * changes of high b-value SI and ADC early during treatment (2weeks after start of therapy; allowed optimal window 10-14 days)
  * treatment follow-up 3 months after initiation of treatment
  of GIST visualized on the WB-DWI as predictor of progression free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Vandecaveye, Prof.Dr., Principal Investigator — University Hospital Gasthuisberg, department of Radiology
Locations (1):
- Radiology Department, Leuven, Leuven, Belgium